CLINICAL TRIAL: NCT05062239
Title: Post-Operative Atrial Fibrillation After Surgical Aortic Valve Replacement and the Influence of Statins - Randomized Controlled Trial
Brief Title: Post-Operative Atrial Fibrillation After Surgical Aortic Valve Replacement and the Influence of Statins
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lars Peter Riber (Other)
Collaborators: Odense Patient Data Explorative Network (Other); GCP-unit at Odense University Hospital (Unknown)
Responsible Party: Sponsor-Investigator, Lars Peter Riber, MD, Associate Professor, Ph.D., DMSc, Odense University Hospital
Organization: Odense University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STARC210421_3; 2021-002210-13 (EudraCT Number)
Record Dates: First submitted 2021-08-19; First posted 2021-09-30 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Postoperative Atrial Fibrillation
MeSH Terms: interventions — Postoperative Period

STUDY DESIGN:
Intervention Model Description: Discontinuous of statin Intervention: Discontinuous of statin, n = 50 Length of preoperative discontinuous: 7 to 14 days prior to surgery Length of postoperative discontinuous: 30 days Control group: continuing medication, n = 50
  No withdrawal study could be found in the literature. We therefore estimate that 100 patients with 50 patients in each group will be enough to observe significant differences, if withdrawal statin should be a clinically manifested issue for the risk of POAF from 36% to 66%.
  Sample size Continuance of statins: 50 Discontinuance of statins: 50
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Continuance (Active Comparator): Continuance prior statin therapy.
  Interventions: Drug: No-intervention.
- Discontinuance (Experimental): Discontinuance prior statin therapy. Duration: From 7 to 14 days prior to surgery until 30 days postoperative
  Interventions: Drug: Discontinuance of treatment with statins 7 to 14 days prior to surgery until 30 days postoperative

INTERVENTIONS:
Drug: Discontinuance of treatment with statins 7 to 14 days prior to surgery until 30 days postoperative — Discontinuance of prior statin therapy
  Arms: Discontinuance
Drug: No-intervention. — Continuance of prior statin therapy
  Arms: Continuance

SUMMARY:
Statins have rapid and significant actions that have potentially important (but not yet proven) implications for postoperative atrial fibrillation and cardiac protection in patients undergoing cardiac surgery.

The focus of this study is, therefore, on patients having surgical aortic valve replacement (with aortotomy) and the development of postoperative atrial fibrillation (POAF).

Our aims are: to investigate the risk of POAF, infection or other complications after SAVR in continuous versus preoperative discontinuous treatment with statins.

The study is a single centre randomized controlled trial with continuance treatment with statin vs. discontinuance (7 to 14 days prior surgery until the 30th post-operative day included), on patients undergoing elective solitary SAVR with bioprosthesis with prior usage of statins the last 3 months and of at least 7 days.

This randomized studies will address 2 separate hypotheses in patients undergoing open heart operation with solitary aortic valve replacement with a bioprosthetic valve that

1. Discontinuation of HMG-CoA reductase inhibitors 7 to 14 days preoperative until 30 days postoperative of AVR in patients with prior use of HMG-CoA reductase inhibitors is not associated with increased early (<30 days) risk of POAF.
2. Discontinuation of HMG-CoA reductase inhibitors 7 to 14 days preoperative until 30 days postoperative of AVR in patients with prior use of HMG-CoA reductase inhibitors is not associated with increased early (<30 days) and intermediate (<1 year) risk of mortality, MI, stroke and rehospitalisation.

DETAILED DESCRIPTION:
Trial Participants:

Enrolment for the study is planned to start February 2022 and continue until 100 patients have been enrolled.

DEFINITION OF POAF:

Postoperative AF (I48) is defined as irregular RR-intervals without a traceable p-wave before each QRS complex during at least 30 seconds or entire 12-lead ECG in symptomatic or asymptomatic patients with no prior history of atrial fibrillation or flutter are considered4. Continuous ECG monitoring (8-lead ward monitor) will recognise AF during the entire hospitalization. Anamnesis, electronic health record (EHR), or confirmatory rhythm strip or 12-lead ECG of AF until 30th postoperative day are also considered.

We will also report the burden of atrial fibrillation, and treatment with a rate controlling drug, antiarrhythmic drug, or electrical cardioversion.

Course of action:

Patients undergoing elective surgical aortic valve replacement with bioprosthesis at the Department of Cardiac Surgery at Odense University Hospital will be offered participation in the study.

Potentially eligible patients will be screened according to inclusion/exclusion criteria at the time after eligibility of surgery. This is assessed at a multidisciplinary team (MDT) conference (with attendance of cardiologist, cardiac surgeons and anaesthesiologist) based on clinical evaluation, echocardiographic ultrasound, coronary angiography and lung function test.

Patients eligible to participate in the study will be presented with the information of the study at the time of their out-patient appointment, according to normal routine at Odense University Hospital. At this appointment the patient receives a physical examination and journal record is obtained by a cardiac surgeon (approximately 7 to 14 days prior to planned surgery).

The study-information will be given by one of the participating doctors, while the patient has been informed of the possibility of bringing an assessor of their choice. The information will be delivered in a quiet room blocked to other appointments in the Department of Cardiothoracic Surgery.

During this meeting the patient will be informed of the purpose of this study and the written patient information will be submitted in detail. Patients will be given as much time as wanted after the oral information has been delivered to decide if they wish to participate in the study. Patients will be offered the possibility to call one of the doctors taking part in this study during this time, in case of additional questions. Subjects can leave the study at any time for any reason if they wish to do so, without any consequences.

Signed informed consent will be provided prior to any research procedures. A subject is registered when signed informed consent has been provided and assigned a subject identification code by the computer-generated code. A subject is randomized when a treatment and a randomisation number has been provided. A subject is considered enrolled in the study once the subject is randomized.

Patient data from EHR will be conducted according to study endpoints after signed informed consent is provided. Signed consent gives sponsor and sponsors representatives

Randomization:

Allocation to a numbered treatment pack (continuance or discontinuance of statin therapy) Randomization scheme will be set-up by OPEN data manager with control for beta-blockers and age (60-65, 66-70, 71-80, >80), and then randomization per se will be executed with the use of REDCap.

The following will be recorded at the day of randomization:

* Conduct information for baseline characteristics
* Transthoracic Echocardiography measurements

Collect baseline blood sample:

• Troponin, CK-MB, Creatinine, CRP

Commence intervention

Perioperative interventions and outcomes from the day of surgery to the day of discharge:

* Duration of aortic cross clamp (ACC), extracorporeal circulation (ECC), ventilatory support, intensive care unit stay period, hospital stay period
* Continue intervention
* Blood samples:

  * Preoperative: Troponin, CK-MB, Creatinine, CRP, Plasma-Atorvastatin
  * Serial troponin and CK-MB levels: (6, 24, 48, and 96 hours after surgery).
  * Creatinine levels: 48 and 96 hours after surgery.
  * CRP levels: 48 and 96 hours after surgery
* Monitor ECG by continuous Holter monitoring to commence as soon as possible after surgery and continue up to post-operative day 5 evening
* Transthoracic Echocardiography on post-operative day 3-5
* Record fluid intake and output during the first 48 hours following surgery based on IV fluids administration, blood transfusion (if applicable), oral/nasogastric intake, and urine plus surgical drain output
* Record intraoperative defibrillation, removal of external pacemaker, new PPM/ICD, vasopressors, blood transfusion, surgical re-exploration, renal replacement therapy, beta-blockers, ACEi/ARB, Amiodarone, Digoxin, Diuretics, Calcium channel blockers, Potassium supplements, NSAIDs or steroids, non-study statin, use of nephrotoxic antibiotics, contrast agents or potassium sparing diuretics (Yes/No)

Assessment at/after discharge from hospital:

* Continue study medications for 30 days after the surgery
* Phone call on the 30th postoperative day to evaluate symptoms of discomfort compatible with atrial fibrillation
* At the end of the study, all excess study medication can be returned at the local drugstore for safe disposal
* Patient data from EHR will be conducted according to study endpoints.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing elective solitary SAVR with bioprosthesis
2. Patients who are in sinus rhythm and not taking any anti-arrhythmic medication, other than beta-adrenergic blocking agents, at the time of surgery
3. In treatment with HMG-CoA reductase inhibitors in the past 3 months and of at least 7 days
4. Age >60 years
5. Willingness and provision of informed consent to be randomized

Exclusion Criteria:

1. Prior history of atrial fibrillation
2. Prior history of cardiac surgery
3. Hepatic dysfunction (Alanin-aminotransferase more than twice the upper limit)
4. Creatinine >200 µmol/L

Ages: 60 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with POAF - In-hospital | In-hospital up to 10 days.
  In-hospital POAF assessed by Holter monitoring.
Number of Participants with POAF - Early | Early (≤30 days) incidence of POAF
  Early assessed by anamnesis and electronic health record (EHR).
Duration of POAF in-hospital | In-hospital
  Duration of POAF monitered with continuous ECG monitoring (eight-- lead ward monitor) up to 24 weeks.

SECONDARY OUTCOMES:
Number of Participants with NOAF | Intermediate (1 year) incidence of NOAF
  NOAF assessed by anamnesis and EHR.
Rate of all-cause mortality - In-hospital | In-hospital up to 10 days.
  Number of deaths in each group.
Rate of all-cause mortality - Early | Early (≤30 days)
  Number of deaths in each group.
Rate of all-cause mortality - intermediate | Intermediate (1 year)
  Number of deaths in each group.
Myocardial injury - Tn | After surgery until discharge up to 10 days
  Injury assessed by serial Troponin measurements. Unit:ng/l
Myocardial injury - CKMB | After surgery until discharge up to 10 days
  Injury assessed by serial CKMB measurements. Unit: μg/l.
Stroke - Early | Early (≤30 days).
  Number of patients with stroke in each group.
Stroke - Intermediate | Intermediate (1 year)
  Number of patients with stroke in each group.
Trans ischemic attack - Early | Early (≤30 days)
  Number of patients with trans ischemic attack in each group.
Trans ischemic attack - Intermediate | Intermediate (1 year)
  Number of patients with trans ischemic attack in each group.
Myocardial infarction - Early | Early (≤30 days)
  Number of patients with Myocardial infarction in each group.
Myocardial infarction - Intermediate | Intermediate (1 year)
  Number of patients with Myocardial infarction in each group.
Permanent pacemaker - Early | Early (≤30 days)
  Number of patients with Permanent pacemaker in each group.
Permanent pacemaker - Intermediate | Intermediate (1 year)
  Number of patients with Permanent pacemaker in each group.
ICD implantation - Early | Early (≤30 days)
  Number of patients with ICD implantation in each group.
ICD implantation - Intermediate | Intermediate (1 year)
  Number of patients with ICD implantation in each group.
Acute kidney injury - Early | Early (≤30 days)
  Number of patients with Acute kidney injury in each group.
LVEF | Before surgery compared with prior to discharge (On the 3rd to 5th postoperative day).
  Describe echocardiography assessed differences in pre and postoperative measurements of LVEF(left ventricular ejection fraction) between groups. Unit: %
Strain | Before surgery compared with prior to discharge (On the 3rd to 5th postoperative day).
  Describe echocardiography assessed differences in pre and postoperative measurements of Strain between groups.Unit: %
TAPSE | Before surgery compared with prior to discharge (On the 3rd to 5th postoperative day).
  Describe echocardiography assessed differences in pre and postoperative measurements of TAPSE (tricuspid annular plane systolic excursion) between groups. Unit: mm
Length of stay on ICU | Day of surgery to the day of discharge from ICU. Up to 52 weeks.
  Length of stay on ICU after surgery. Unit: Days
Length of stay in hospital | Day of surgery to the day of discharge from the hospital. Up to 52 weeks.
  Length of stay in hospital after surgery. Unit: Days

CONTACTS AND LOCATIONS:
Locations (1):
- Odense University Hospital, Odense, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Data will be available in anonymized form in accordance with GDPR upon reasonable request.
  Rules for external researchers to apply for and access data will be laid out towards the end of the study.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: TBA
Access Criteria: TBA

REFERENCES:
- [Background] LaPar DJ, Crosby IK, Rich JB, Fonner E Jr, Kron IL, Ailawadi G, Speir AM; Investigators for Virginia Cardiac Surgery Quality Initiative. A contemporary cost analysis of postoperative morbidity after coronary artery bypass grafting with and without concomitant aortic valve replacement to improve patient quality and cost-effective care. Ann Thorac Surg. 2013 Nov;96(5):1621-7. doi: 10.1016/j.athoracsur.2013.05.050. Epub 2013 Aug 21. PMID 23972932
- [Background] Brown JM, O'Brien SM, Wu C, Sikora JA, Griffith BP, Gammie JS. Isolated aortic valve replacement in North America comprising 108,687 patients in 10 years: changes in risks, valve types, and outcomes in the Society of Thoracic Surgeons National Database. J Thorac Cardiovasc Surg. 2009 Jan;137(1):82-90. doi: 10.1016/j.jtcvs.2008.08.015. PMID 19154908
- [Background] Maesen B, Nijs J, Maessen J, Allessie M, Schotten U. Post-operative atrial fibrillation: a maze of mechanisms. Europace. 2012 Feb;14(2):159-74. doi: 10.1093/europace/eur208. Epub 2011 Aug 6. PMID 21821851
- [Background] Hindricks G, Potpara T, Dagres N, Arbelo E, Bax JJ, Blomstrom-Lundqvist C, Boriani G, Castella M, Dan GA, Dilaveris PE, Fauchier L, Filippatos G, Kalman JM, La Meir M, Lane DA, Lebeau JP, Lettino M, Lip GYH, Pinto FJ, Thomas GN, Valgimigli M, Van Gelder IC, Van Putte BP, Watkins CL; ESC Scientific Document Group. 2020 ESC Guidelines for the diagnosis and management of atrial fibrillation developed in collaboration with the European Association for Cardio-Thoracic Surgery (EACTS): The Task Force for the diagnosis and management of atrial fibrillation of the European Society of Cardiology (ESC) Developed with the special contribution of the European Heart Rhythm Association (EHRA) of the ESC. Eur Heart J. 2021 Feb 1;42(5):373-498. doi: 10.1093/eurheartj/ehaa612. No abstract available. PMID 32860505
- [Background] Arsenault KA, Yusuf AM, Crystal E, Healey JS, Morillo CA, Nair GM, Whitlock RP. Interventions for preventing post-operative atrial fibrillation in patients undergoing heart surgery. Cochrane Database Syst Rev. 2013 Jan 31;2013(1):CD003611. doi: 10.1002/14651858.CD003611.pub3. PMID 23440790
- [Background] AlTurki A, Marafi M, Proietti R, Cardinale D, Blackwell R, Dorian P, Bessissow A, Vieira L, Greiss I, Essebag V, Healey JS, Huynh T. Major Adverse Cardiovascular Events Associated With Postoperative Atrial Fibrillation After Noncardiac Surgery: A Systematic Review and Meta-Analysis. Circ Arrhythm Electrophysiol. 2020 Jan;13(1):e007437. doi: 10.1161/CIRCEP.119.007437. Epub 2020 Jan 16. PMID 31944855
- [Background] Dobrev D, Aguilar M, Heijman J, Guichard JB, Nattel S. Postoperative atrial fibrillation: mechanisms, manifestations and management. Nat Rev Cardiol. 2019 Jul;16(7):417-436. doi: 10.1038/s41569-019-0166-5. PMID 30792496
- [Background] Greenberg JW, Lancaster TS, Schuessler RB, Melby SJ. Postoperative atrial fibrillation following cardiac surgery: a persistent complication. Eur J Cardiothorac Surg. 2017 Oct 1;52(4):665-672. doi: 10.1093/ejcts/ezx039. PMID 28369234
- [Background] Aguilar M, Dobrev D, Nattel S. Postoperative Atrial Fibrillation: Features, Mechanisms, and Clinical Management. Card Electrophysiol Clin. 2021 Mar;13(1):123-132. doi: 10.1016/j.ccep.2020.11.010. PMID 33516390
- [Background] Kim YM, Kattach H, Ratnatunga C, Pillai R, Channon KM, Casadei B. Association of atrial nicotinamide adenine dinucleotide phosphate oxidase activity with the development of atrial fibrillation after cardiac surgery. J Am Coll Cardiol. 2008 Jan 1;51(1):68-74. doi: 10.1016/j.jacc.2007.07.085. PMID 18174039
- [Background] Antoniades C, Demosthenous M, Reilly S, Margaritis M, Zhang MH, Antonopoulos A, Marinou K, Nahar K, Jayaram R, Tousoulis D, Bakogiannis C, Sayeed R, Triantafyllou C, Koumallos N, Psarros C, Miliou A, Stefanadis C, Channon KM, Casadei B. Myocardial redox state predicts in-hospital clinical outcome after cardiac surgery effects of short-term pre-operative statin treatment. J Am Coll Cardiol. 2012 Jan 3;59(1):60-70. doi: 10.1016/j.jacc.2011.08.062. PMID 22192670
- [Background] Scott L Jr, Li N, Dobrev D. Role of inflammatory signaling in atrial fibrillation. Int J Cardiol. 2019 Jul 15;287:195-200. doi: 10.1016/j.ijcard.2018.10.020. Epub 2018 Oct 4. PMID 30316645
- [Background] Wong CX, Ganesan AN, Selvanayagam JB. Epicardial fat and atrial fibrillation: current evidence, potential mechanisms, clinical implications, and future directions. Eur Heart J. 2017 May 1;38(17):1294-1302. doi: 10.1093/eurheartj/ehw045. PMID 26935271
- [Background] Halonen J, Halonen P, Jarvinen O, Taskinen P, Auvinen T, Tarkka M, Hippelainen M, Juvonen T, Hartikainen J, Hakala T. Corticosteroids for the prevention of atrial fibrillation after cardiac surgery: a randomized controlled trial. JAMA. 2007 Apr 11;297(14):1562-7. doi: 10.1001/jama.297.14.1562. PMID 17426275
- [Background] Zheng Z, Jayaram R, Jiang L, Emberson J, Zhao Y, Li Q, Du J, Guarguagli S, Hill M, Chen Z, Collins R, Casadei B. Perioperative Rosuvastatin in Cardiac Surgery. N Engl J Med. 2016 May 5;374(18):1744-53. doi: 10.1056/NEJMoa1507750. PMID 27144849
- [Background] Pinho-Gomes AC, Reilly S, Brandes RP, Casadei B. Targeting inflammation and oxidative stress in atrial fibrillation: role of 3-hydroxy-3-methylglutaryl-coenzyme a reductase inhibition with statins. Antioxid Redox Signal. 2014 Mar 10;20(8):1268-85. doi: 10.1089/ars.2013.5542. Epub 2013 Oct 19. PMID 23924190
- [Background] Oesterle A, Laufs U, Liao JK. Pleiotropic Effects of Statins on the Cardiovascular System. Circ Res. 2017 Jan 6;120(1):229-243. doi: 10.1161/CIRCRESAHA.116.308537. PMID 28057795
- [Background] Thiago L, Tsuji SR, Nyong J, Puga ME, Gois AF, Macedo CR, Valente O, Atallah AN. Statins for aortic valve stenosis. Cochrane Database Syst Rev. 2016 Sep 5;9(9):CD009571. doi: 10.1002/14651858.CD009571.pub2. PMID 27594276
- [Background] Davignon J. Beneficial cardiovascular pleiotropic effects of statins. Circulation. 2004 Jun 15;109(23 Suppl 1):III39-43. doi: 10.1161/01.CIR.0000131517.20177.5a. PMID 15198965
- [Background] Blanco-Colio LM, Tunon J, Martin-Ventura JL, Egido J. Anti-inflammatory and immunomodulatory effects of statins. Kidney Int. 2003 Jan;63(1):12-23. doi: 10.1046/j.1523-1755.2003.00744.x. PMID 12472764
- [Background] Fauchier L, Clementy N, Babuty D. Statin therapy and atrial fibrillation: systematic review and updated meta-analysis of published randomized controlled trials. Curr Opin Cardiol. 2013 Jan;28(1):7-18. doi: 10.1097/HCO.0b013e32835b0956. PMID 23160338
- [Background] Fang WT, Li HJ, Zhang H, Jiang S. The role of statin therapy in the prevention of atrial fibrillation: a meta-analysis of randomized controlled trials. Br J Clin Pharmacol. 2012 Nov;74(5):744-56. doi: 10.1111/j.1365-2125.2012.04258.x. PMID 22376147
- [Background] Mannacio VA, Iorio D, De Amicis V, Di Lello F, Musumeci F. Effect of rosuvastatin pretreatment on myocardial damage after coronary surgery: a randomized trial. J Thorac Cardiovasc Surg. 2008 Dec;136(6):1541-8. doi: 10.1016/j.jtcvs.2008.06.038. Epub 2008 Aug 15. PMID 19114204
- [Background] Almansob MA, Xu B, Zhou L, Hu XX, Chen W, Chang FJ, Ci HB, Yao JP, Xu YQ, Yao FJ, Liu DH, Zhang WB, Tang BY, Wang ZP, Ou JS. Simvastatin reduces myocardial injury undergoing noncoronary artery cardiac surgery: a randomized controlled trial. Arterioscler Thromb Vasc Biol. 2012 Sep;32(9):2304-13. doi: 10.1161/ATVBAHA.112.252098. Epub 2012 Jul 12. PMID 22796581
- [Background] Kuhn EW, Liakopoulos OJ, Stange S, Deppe AC, Slottosch I, Choi YH, Wahlers T. Preoperative statin therapy in cardiac surgery: a meta-analysis of 90,000 patients. Eur J Cardiothorac Surg. 2014 Jan;45(1):17-26; discussion 26. doi: 10.1093/ejcts/ezt181. Epub 2013 Apr 5. PMID 23562936
- [Background] Kuhn EW, Slottosch I, Wahlers T, Liakopoulos OJ. Preoperative statin therapy for patients undergoing cardiac surgery. Cochrane Database Syst Rev. 2015 Aug 13;(8):CD008493. doi: 10.1002/14651858.CD008493.pub3. PMID 26270008
- [Background] Patti G, Chello M, Candura D, Pasceri V, D'Ambrosio A, Covino E, Di Sciascio G. Randomized trial of atorvastatin for reduction of postoperative atrial fibrillation in patients undergoing cardiac surgery: results of the ARMYDA-3 (Atorvastatin for Reduction of MYocardial Dysrhythmia After cardiac surgery) study. Circulation. 2006 Oct 3;114(14):1455-61. doi: 10.1161/CIRCULATIONAHA.106.621763. Epub 2006 Sep 25. PMID 17000910
- [Background] Ji Q, Mei Y, Wang X, Sun Y, Feng J, Cai J, Xie S, Chi L. Effect of preoperative atorvastatin therapy on atrial fibrillation following off-pump coronary artery bypass grafting. Circ J. 2009 Dec;73(12):2244-9. doi: 10.1253/circj.cj-09-0352. Epub 2009 Oct 13. PMID 19822977
- [Background] Sun Y, Ji Q, Mei Y, Wang X, Feng J, Cai J, Chi L. Role of preoperative atorvastatin administration in protection against postoperative atrial fibrillation following conventional coronary artery bypass grafting. Int Heart J. 2011;52(1):7-11. doi: 10.1536/ihj.52.7. PMID 21321461
- [Background] Zhang L, Zhang S, Jiang H, Sun A, Wang Y, Zou Y, Ge J, Chen H. Effects of statin therapy on inflammatory markers in chronic heart failure: a meta-analysis of randomized controlled trials. Arch Med Res. 2010 Aug;41(6):464-71. doi: 10.1016/j.arcmed.2010.08.009. PMID 21044751
- [Background] Vukovic PM, Maravic-Stojkovic VR, Peric MS, Jovic MDj, Cirkovic MV, Gradinac SDj, Djukanovic BP, Milojevic PS. Steroids and statins: an old and a new anti-inflammatory strategy compared. Perfusion. 2011 Jan;26(1):31-7. doi: 10.1177/0267659110385607. Epub 2010 Oct 4. PMID 20921085
- [Background] Antoniades C, Bakogiannis C, Tousoulis D, Reilly S, Zhang MH, Paschalis A, Antonopoulos AS, Demosthenous M, Miliou A, Psarros C, Marinou K, Sfyras N, Economopoulos G, Casadei B, Channon KM, Stefanadis C. Preoperative atorvastatin treatment in CABG patients rapidly improves vein graft redox state by inhibition of Rac1 and NADPH-oxidase activity. Circulation. 2010 Sep 14;122(11 Suppl):S66-73. doi: 10.1161/CIRCULATIONAHA.109.927376. PMID 20837928
- [Background] Song YB, On YK, Kim JH, Shin DH, Kim JS, Sung J, Lee SH, Kim WS, Lee YT. The effects of atorvastatin on the occurrence of postoperative atrial fibrillation after off-pump coronary artery bypass grafting surgery. Am Heart J. 2008 Aug;156(2):373.e9-16. doi: 10.1016/j.ahj.2008.04.020. Epub 2008 Jun 17. PMID 18657672
- [Background] Chello M, Patti G, Candura D, Mastrobuoni S, Di Sciascio G, Agro F, Carassiti M, Covino E. Effects of atorvastatin on systemic inflammatory response after coronary bypass surgery. Crit Care Med. 2006 Mar;34(3):660-7. doi: 10.1097/01.CCM.0000201407.89977.EA. PMID 16505650
- [Background] Macin SM, Perna ER, Farias EF, Franciosi V, Cialzeta JR, Brizuela M, Medina F, Tajer C, Doval H, Badaracco R. Atorvastatin has an important acute anti-inflammatory effect in patients with acute coronary syndrome: results of a randomized, double-blind, placebo-controlled study. Am Heart J. 2005 Mar;149(3):451-7. doi: 10.1016/j.ahj.2004.07.041. PMID 15864233
- [Background] Ridker PM, Cannon CP, Morrow D, Rifai N, Rose LM, McCabe CH, Pfeffer MA, Braunwald E; Pravastatin or Atorvastatin Evaluation and Infection Therapy-Thrombolysis in Myocardial Infarction 22 (PROVE IT-TIMI 22) Investigators. C-reactive protein levels and outcomes after statin therapy. N Engl J Med. 2005 Jan 6;352(1):20-8. doi: 10.1056/NEJMoa042378. PMID 15635109
- [Background] Hashemzadeh K, Dehdilani M, Dehdilani M. Postoperative Atrial Fibrillation following Open Cardiac Surgery: Predisposing Factors and Complications. J Cardiovasc Thorac Res. 2013;5(3):101-7. doi: 10.5681/jcvtr.2013.022. Epub 2013 Oct 5. PMID 24252985
- [Background] Fragao-Marques M, Mancio J, Oliveira J, Falcao-Pires I, Leite-Moreira A. Gender Differences in Predictors and Long-Term Mortality of New-Onset Postoperative Atrial Fibrillation Following Isolated Aortic Valve Replacement Surgery. Ann Thorac Cardiovasc Surg. 2020 Dec 20;26(6):342-351. doi: 10.5761/atcs.oa.19-00314. Epub 2020 Apr 28. PMID 32350163
- [Background] Turagam MK, Downey FX, Kress DC, Sra J, Tajik AJ, Jahangir A. Pharmacological strategies for prevention of postoperative atrial fibrillation. Expert Rev Clin Pharmacol. 2015 Mar;8(2):233-50. doi: 10.1586/17512433.2015.1018182. PMID 25697411
- [Background] Zebis LR, Christensen TD, Thomsen HF, Mikkelsen MM, Folkersen L, Sorensen HT, Hjortdal VE. Practical regimen for amiodarone use in preventing postoperative atrial fibrillation. Ann Thorac Surg. 2007 Apr;83(4):1326-31. doi: 10.1016/j.athoracsur.2006.09.096. PMID 17383335
- [Background] Crystal E, Connolly SJ, Sleik K, Ginger TJ, Yusuf S. Interventions on prevention of postoperative atrial fibrillation in patients undergoing heart surgery: a meta-analysis. Circulation. 2002 Jul 2;106(1):75-80. doi: 10.1161/01.cir.0000021113.44111.3e. PMID 12093773
- [Background] Taira CA, Opezzo JA, Mayer MA, Hocht C. Cardiovascular drugs inducing QT prolongation: facts and evidence. Curr Drug Saf. 2010 Jan;5(1):65-72. doi: 10.2174/157488610789869229. PMID 20210721
- [Background] Taylor F, Huffman MD, Macedo AF, Moore TH, Burke M, Davey Smith G, Ward K, Ebrahim S. Statins for the primary prevention of cardiovascular disease. Cochrane Database Syst Rev. 2013 Jan 31;2013(1):CD004816. doi: 10.1002/14651858.CD004816.pub5. PMID 23440795
- [Background] Adams SP, Tsang M, Wright JM. Lipid-lowering efficacy of atorvastatin. Cochrane Database Syst Rev. 2015 Mar 12;2015(3):CD008226. doi: 10.1002/14651858.CD008226.pub3. PMID 25760954
- [Background] Newman C, Tsai J, Szarek M, Luo D, Gibson E. Comparative safety of atorvastatin 80 mg versus 10 mg derived from analysis of 49 completed trials in 14,236 patients. Am J Cardiol. 2006 Jan 1;97(1):61-7. doi: 10.1016/j.amjcard.2005.07.108. Epub 2005 Nov 15. PMID 16377285
- [Background] Cholesterol Treatment Trialists' (CTT) Collaboration; Baigent C, Blackwell L, Emberson J, Holland LE, Reith C, Bhala N, Peto R, Barnes EH, Keech A, Simes J, Collins R. Efficacy and safety of more intensive lowering of LDL cholesterol: a meta-analysis of data from 170,000 participants in 26 randomised trials. Lancet. 2010 Nov 13;376(9753):1670-81. doi: 10.1016/S0140-6736(10)61350-5. Epub 2010 Nov 8. PMID 21067804
- [Background] Hansen MR, Hrobjartsson A, Pottegard A, Damkier P, Madsen KG, Pareek M, Olesen M, Hallas J. Postponement of cardiovascular outcomes by statin use: A systematic review and meta-analysis of randomized clinical trials. Basic Clin Pharmacol Toxicol. 2021 Feb;128(2):286-296. doi: 10.1111/bcpt.13485. Epub 2020 Oct 8. PMID 32896109